CLINICAL TRIAL: NCT03018067
Title: A Single-Blind, Placebo-Controlled Study Evaluating the Onset-of-Action, Safety, and Efficacy of RDX227675 for the Treatment of Hyperkalemia
Brief Title: A Study Evaluating the Onset-of-Action, Safety, and Efficacy of RDX227675 for the Treatment of Hyperkalemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor stopped program]
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDX227675-201
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Microcrystalline Cellulose (MCC), 2 g qd. Subjects assigned to the Placebo group will be randomly assigned in a 1:1:1 ratio to receive either one, two, or three bottles of drug per day.
  Interventions: Drug: Placebo
- 10 g qd (Experimental): RDX227675, 10 g qd
  Interventions: Drug: RDX227675
- 20 g qd (Experimental): RDX227675, 20 g qd
  Interventions: Drug: RDX227675
- 30 g qd (Experimental): RDX227675, 30 g qd
  Interventions: Drug: RDX227675

INTERVENTIONS:
Drug: RDX227675
  Arms: 10 g qd; 20 g qd; 30 g qd
Drug: Placebo
  Arms: Placebo

SUMMARY:
This phase 2, single-blind, placebo-controlled study will evaluate the onset-of-action, safety, and efficacy of RDX227675 for the treatment of hyperkalemia. Subjects who qualify are randomized into one of four treatment groups: Group 1 (Placebo qd), Group 2 (RDX227675 10 g qd), Group 3 (RDX227675 20 g qd), Group 4 (RDX227675 30 g qd).

DETAILED DESCRIPTION:
The study consists of a screening visit, a 7-day treatment period, and a 7-day treatment-free follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years old, inclusive
* Two consecutive i-STAT K values ≥ 5.5 to < 6.5 mmol/L, measured a minimum of 60-minutes apart within 1 day of first RDX227675 dose on Day 1 (prior to randomization)
* i-STAT K value ≥ 5.5 to < 6.5 mmol/L on Day 1 (prior to randomization)
* Ability to have repeated blood draws or effective venous catheterization
* Females of child bearing potential must have negative urine pregnancy test on Day 1 (prior to randomization)
* Females but be non-pregnant, non-lactating, and either be post-menopausal for at least 12 months, have documentation of irreversible surgical sterilization, or confirm the use of one of the acceptable contraceptive methods
* Males must agree to use an appropriate method of contraception or have documented surgical sterilization

Exclusion Criteria:

* Pseudohyperkalemia signs and symptoms
* Treatment with K lowering drugs, within 7 days prior to randomization
* Uncontrolled Type 2 diabetes, as defined as most recent historical HbA1c > 10%, or hospitalization to treat hyper- or hypo-glycemia in the past 3 months
* Diabetic ketoacidosis
* Known hypersensitivity to polystyrene sulfonate
* Significant cardiovascular or cerebrovascular events in the past 2 months
* Severe heart failure, defined as NYHA (New York Heart Association) class IV or hospitalization to treat heart failure in previous 3 months
* History of bowel obstruction, swallowing disorders, severe gastrointestinal disorders, or major gastrointestinal surgery
* Major psychiatric disorder (DSM-III-R or DSM-IV) including major depression or other psychoses that has required hospitalization in the last 3 years. History of attempted suicide or uncontrolled bipolar disorder.
* Use of an investigational product within 30 days prior to Screening

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Exponential Rate of Change in Serum Potassium from Baseline | 48 hours
  Onset of Action

SECONDARY OUTCOMES:
Change in Serum Potassium Levels | 7 days
Incidence of Treatment - Emergent Adverse Events [Safety and Tolerability] | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Chair — Ardelyx, Inc.
Locations (1):
- Capital Nephrology Associates, PA, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No